CLINICAL TRIAL: NCT00663429
Title: A Phase II Open-Label Extension Study of the Safety and Efficacy of Atiprimod Treatment for Patients With Low to Intermediate Grade Neuroendocrine Carcinoma
Brief Title: Extension Study of the Safety and Efficacy of Atiprimod Treatment in Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Callisto Pharmaceuticals (Industry)
Responsible Party: Gary S. Jacob, PhD Chief Executive Officer, Callisto Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-AT202-07
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2009-01

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — azaspirane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atiprimod — Oral, 14 days on / 14 days off; 30mg capsules

SUMMARY:
This study is an extension study to the Callisto protocol CP-106. Subjects must have completed all 12 treatment cycles of CP-106 without disease progression as per RECIST criteria,to be eligible to to be enrolled in this study. This study will evaluate the safety and efficacy of atiprimod treatment in patients with low to intermediate grade neuroendocrine carcinoma who have metastatic or unresectable local-regional cancer and who have either symptoms (diarrhea, flushing and/or wheezing) despite standard therapy (octreotide) or progression of neuroendocrine tumor(s).

DETAILED DESCRIPTION:
For carcinoid, despite the many cytotoxic chemotherapy trials that have been conducted, no regimen has demonstrated a response rate of more than 20% using the criterion of a 50% reduction of bidimensionally measurable disease. In the more recently reported ECOG phase III study of chemotherapy in carcinoid tumors (E1281), patients were randomly assigned to treatment with 5-fluorouracil (5FU) plus doxorubicin or 5FU plus streptozocin. The median progression free survival durations were disappointing. They were 4.5 months in the 5FU plus doxorubicin arm and 5.3 months in the 5FU plus streptozocin arm. Overall survival durations recorded in the trial were also suboptimal at 15 and 24 months respectively. There is no clear survival benefit for cytotoxic chemotherapy.

This is a phase II, multi-center, open-label extension study of the safety and efficacy of atiprimod treatment in patients with low to intermediate grade neuroendocrine carcinoma who have metastatic or unresectable local-regional cancer and who have either symptoms (diarrhea, flushing and/or wheezing) despite standard therapy (octreotide) or progression of neuroendocrine tumor(s) (defined as the appearance of one or more new lesions or a 20% increase in the sum of the longest diameter of target lesions during the 6 months prior to enrollment in CP-106). Atiprimod will be administered orally as a single daily dose of 60 mg/day for 14 days, followed by a 14-day treatment-free period (i.e., 1 treatment cycle = 28 days).

ELIGIBILITY:
Inclusion Criteria:

1. Subject was enrolled in Protocol No. CP-106 and successfully completed 12 treatment cycles.
2. Subject must have been classified as a responder at the time of completion of Protocol No. CP-106 [i.e., SD or better per RECIST Committee criteria or stable symptoms or better (defined as an average daily frequency of bowel movements, flushing episodes and/or wheezing episodes that is the same as or less than the average daily frequency of bowel movements, flushing episodes and/or wheezing episodes recorded during the 14-day screening period prior to enrollment in Protocol No. CP-106)].
3. Subject must understand and voluntarily sign the informed consent document.
4. Subject must have adequate organ function defined as follows: Absolute granulocyte count (AGC) >1,500/mm3, hemoglobin >8 g/dl, platelets >100,000/mm3, serum bilirubin <1.5 x upper limit of normal (ULN), serum creatinine <1.5 mg/dL, SGOT ≤Grade 1 per NCI CTCAE, SGPT ≤Grade 1 per NCI CTCAE.
5. Women of child bearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable or implantable hormonal contraceptive; tubal ligation; intra-uterine devices; barrier contraceptive with spermicide; or vasectomized partner).

Exclusion Criteria:

1. Subject who was enrolled in Protocol No. CP-106 and who did not successfully complete 12 treatment cycles.
2. If WCBP, pregnant, lactating or not using adequate contraception.
3. Clinically relevant active infection or serious co-morbid medical conditions that are uncontrolled or whose control may be jeopardized by atiprimod treatment.
4. Psychiatric disorders rendering subjects incapable of complying with the requirements of the protocol.
5. Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
6. As atiprimod is a potent inhibitor of CYP2D6, the use of drugs that are substrates of CYP2D6 (e.g. beta blockers, antidepressants, and antipsychotic;) will not be allowed while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Reduction of symptoms (diarrhea, flushing and/or wheezing) | 1 year
Progression of neuroendocrine tumor(s) | 1 year

SECONDARY OUTCOMES:
Adverse Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Jacob, PhD, Study Director — Callisto Pharmaceuticals
Locations (2):
- United States (2):
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Mount Sinai Medical Center, New York, New York